CLINICAL TRIAL: NCT05450302
Title: To Assess the Predictive Value of High Frequency Algorithm of PURE EP for Low Amplitude Signal Detection
Brief Title: Assessing the Predictive Value of High Frequency Algorithm of PURE EP for Low Amplitude Signal Detection
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kansas City Heart Rhythm Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KCHRRF-PURE EP-0011
Record Dates: First submitted 2022-06-30; First posted 2022-07-08 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2022-06

CONDITIONS: Cardiac Arrhythmias
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PURE EP: All patients from January 2022 till June 2022 in whom PURE EP was used at the Kansas City Heart Rhythm Institute, Overland Park, Kansas
  Interventions: Other: PURE EP (Observational Study)

INTERVENTIONS:
Other: PURE EP (Observational Study) — This is an observational study. No interventions involved in this study.

SUMMARY:
Prior multicenter study demonstrated superiority of PURE EP to conventional mapping. This superiority was seen when comparing small, fractionated signals of interest, near-field vs far-field distinction, and general signal quality (2). Hence, investigators propose a retrospective study to assess the predictive value of high frequency algorithm (HFA) for identifying local physiologic signal under 0.3 mV distinctive of noise.

DETAILED DESCRIPTION:
Accurate interpretation of intracardiac EGMs remains essential to the field of electrophysiology (EP). Conventional Electro-anatomical mapping systems (EAMs) have made significant improvements in EGM quality and noise reduction since their emergence, however their use of variable gain amplifiers and high/low pass filters, often provide visualization of low amplitude signals that lead to saturation artifact or necessitate signal clipping.

PURE EPTM (BioSig Technologies, Inc., Westport, CT, USA), in contrast does provide the ability to record this unaltered signal with more customizable display options. Their proprietary amplifier and high-resolution analog-digital converters with Radiofrequency (RF) suppression eliminates the need for gain switching, optimizing resolution of the full range of input signals (1).

Prior multicenter study demonstrated superiority of PURE EP to conventional mapping. This superiority was seen when comparing small, fractionated signals of interest, near-field vs far-field distinction, and general signal quality (2). Hence, investigators propose a retrospective study to assess the predictive value of high frequency algorithm (HFA) for identifying local physiologic signal under 0.3 mV distinctive of noise.

ELIGIBILITY:
Inclusion Criteria:

All patients (male + Female) with age > 18 years from January 2022 till June 2022 will be included in the study.

Exclusion Criteria:

All patients in which PURE EP was not used from January 2022 till June 2022.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from January 2022 till June 2022 in whom PURE EP was used at the Kansas City Heart Rhythm Institute, Overland Park, Kansas will be included in the study.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Predictive value of High Frequency Algorithm - for signals under 0.3mV distinctive of noise | 1/1/2022 - 6/30/2022
  Validate the predictive value of High Frequency Algorithm (HFA) for identifying local physiologic signals under 0.3mV distinctive of noise.
Predictive value of High Frequency Algorithm - for signals under 0.1mV distinctive of noise | 1/1/2022 - 6/30/2022
  Validate the predictive value of High Frequency Algorithm (HFA) for identifying local physiologic signals under 0.1mV distinctive of noise
Sensitivity and specificity | 1/1/2022 - 6/30/2022
  Percen of sensitivity and specificity of predicting a small physiologic signal distinctive from noise

SECONDARY OUTCOMES:
Bipolar amplitude | 1/1/2022 - 6/30/2022
  The measurement tool, specifically within PURE EP, called "Horizontal Caliper Mode" similar to that of recording and mapping systems, will measure the millivolt peak-to-peak amplitude of the bipolar signal, which is identified by its electrode numbers.
Channel of the Bipolar | 1/1/2022 - 6/30/2022
  It depends on which channel has the low amplitude signal and it may change based on the signal. It is measured by "Horizontal Caliper Mode '' in millivolts in the PURE EP program.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Kansas City Heart Rhythm Institute, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Padmanabhan D, Foxall T, Drakulic B, Witt C, Killu A, Naksuk N, Sugrue A, Venkatachalam KL, Asirvatham S. Initial Experience with the BioSig PURE EP Signal Recording System: An Animal Laboratory Experience. J Innov Card Rhythm Manag. 2017 Apr 15;8(4):2690-2699. doi: 10.19102/icrm.2017.080407. eCollection 2017 Apr. PMID 32494447
- [Background] Al-Ahmad A, Knight B, Tzou W, Schaller R, Yasin O, Padmanabhan D, Zagrodzky J, Bassiouny M, Burkhardt JD, Gallinghouse GJ, Mansour M, McLeod C, Natale A. Evaluation of a novel cardiac signal processing system for electrophysiology procedures: The PURE EP 2.0 study. J Cardiovasc Electrophysiol. 2021 Nov;32(11):2915-2922. doi: 10.1111/jce.15250. Epub 2021 Oct 1. PMID 34554634